CLINICAL TRIAL: NCT05548829
Title: Covid Response Study (COVRES): A Northern Ireland Population Study of SARS-CoV-2 Prevalence, Predisposing Factors, and Pathology
Brief Title: COVID RESPONSE STUDY (COVRES)
Acronym: COVRES
Status: Completed | Type: Observational
Sponsor: University of Ulster (Other)
Collaborators: University of Dublin, Trinity College (Other); Western Health and Social Care Trust (Other)
Responsible Party: Sponsor
Other Study IDs: COVRES_Ver13; COVRES2 (Other: Ulster University)
Record Dates: First submitted 2022-09-07; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
Keywords: Covid-19; Biomarkers; Severity; Genomics
MeSH Terms: conditions — COVID-19 | interventions — Patient Acuity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — COVRES1 (Case n=519); retrospective cohort. Hospitalised and Non-Hospitalised COVID-19 patients. Collecting DNA and RNA from saliva and Whole blood samples.
  COVRES2 (Case n=42); prospective cohort. Hospitalised and Non-Hospitalised COVID-19 patients. Three and six month follow up. Collecting DNA and RNA from saliva and Whole blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Non-hospitalised Covid-19 patients (mild infection): COVRES1, retrospective recuitment from public advertisment, attended CTRIC or home visits. Obtained saliva and whole blood samples for DNA and RNA extraction.
- Hospitalised Covid-19 patients (severe infection): COVRES1, retrospective recuitment from secondary care, attended wards. Obtained saliva and whole blood samples for DNA and RNA extraction.
  Interventions: Biological: Disease severity
- Non-hospitalised Covid-19 patients (mild infection) 3 month follow up: COVRES2, prospective recuitment, attended CTRIC or home visits. Obtained saliva and whole blood samples for DNA and RNA extraction.
- Hospitalised Covid-19 patients (severe infection) 3 month follow up: COVRES2, prospective recuitment, attended CTRIC or home visits. Obtained saliva and whole blood samples for DNA and RNA extraction.
  Interventions: Biological: Disease severity
- Non-hospitalised Covid-19 patients (mild infection) 6 month follow up: COVRES2, prospective recuitment, attended CTRIC or home visits. Obtained saliva and whole blood samples for DNA and RNA extraction.
- Hospitalised Covid-19 patients (severe infection) 6 month follow up: COVRES2, prospective recuitment, attended CTRIC or home visits. Obtained saliva and whole blood samples for DNA and RNA extraction.
  Interventions: Biological: Disease severity

INTERVENTIONS:
Biological: Disease severity — Observational, based on biological outcome of Covid-19 infeection. Comparing pheripheral biomakers of Covid-19 patients admitted to hospital due to infection versus Covid-19 patients that recovered at home.
  Groups: Hospitalised Covid-19 patients (severe infection); Hospitalised Covid-19 patients (severe infection) 3 month follow up; Hospitalised Covid-19 patients (severe infection) 6 month follow up

SUMMARY:
This study will undertake recruitment of Covid-19 positive hospitalised and non-hospitalised and nursing home patients, hospital and nursing home staff, for whole genome sequencing, human host genomic analyses and viral genomic analyses. This research study will take place across three trust areas in Northern Ireland.

DETAILED DESCRIPTION:
Hospital and nursing home patient recruitment:

COVID-19 positive/ SARS-CoV-2 inpatients and non-hospitalised patients (n = 700) aged 18 years and over tested at the WHSCT, BHSCT and SHSCT and have been admitted to COVID-19/ SARS-CoV-2 hospital wards (including from the Intensive Care Units) or out-patient and residents of trust affiliated nursing homes will initially be approached by their clinician, senior nurse or an NICRN research nurse. Investigators will speak to the patient(s) about the study and if the patient is interested, verbal consent will be gained for the researcher to follow up with a Participant Information sheet (PIS) (appendix 6). Those interested patients fulfilling the inclusion criteria can then speak directly face to face (whereby the nurse will arrange a convenient time for researcher to visit the patient) to the researchers, the study will be discussed in detail and any issues will be addressed. If participants are still interested in participating, written informed consent (appendix 7) will be obtained by the researcher(s) prior to enrolment on the study.

In the case of those ALC, and where a family member is not available to act as a nominated person the research team in conjunction with the PI will identify a nominated person who is unrelated to the conduct of the research and willing to provide a declaration for this study. The nominated person will always be a member of the nursing staff or the management team and part of the wider multi-disciplinary team within the hospital ward or nursing home facility of the individual lacking capacity. The nominated person will also be provided with an invitation letter and PIS (appendix 13) and any queries answered, the nominated person can then contact the research team if it is thought the potential participant would have been interested in this research. The potential participant will not be enrolled on the study until full informed consent (appendix 14) has been given by the nominated person. This will still apply at all time points for those individuals who are unlikely to regain capacity and for those patients in hospital who are sedated/ventilated due to their COVID-19 symptoms, who may regain capacity. For those patients, capacity will always be assessed by a member of their direct clinical care team, the nurse in charge/manager in the nursing home and the PI at each hospital site who will be the consultant on or linked to the COVID ward (The person assessing capacity will be recorded at all time points and a record kept). For those that regain capacity during the duration of this research, a participant information sheet will be provided (appendix 4) to read and consent (appendix 5) will be sought if there are wishes to proceed with the study. If participants do not wish to continue, the option will be provided for any samples and data to be withdrawn and destroyed.

Sample Collection: Once informed consent has been obtained each participant will provide (i) one 30 ml whole blood sample, a saliva sample (~4ml) and one set of up to five 20ul dried blood spots (DBS; equivalent to five finger lancet blood droplets) and a lateral flow assay for COVID-19 antibodies performed at recruitment (between 0 and 10 days of symptom onset), (ii) again between 14-28 days after symptom onset (iii) again samples will be collected only if pneumonia occurs during episode (usually only in severe symptom cases) (iv) In addition, where possible samples will be collected at post 3 months, 6 months, 12 months and 18 months post symptom onset, the latter sample collections will take place at an agreed convenient time and place.

Hospital and nursing home staff recruitment:

All HSC employees aged 18 years and over, employed within facilities at the WHSCT, BHSCT and the SHSCT and trust affiliated nursing homes within the trust areas (n = 500) are eligible to participate in this research. Trust/nursing home wide emails with an attached PIS explaining the study (appendix 6) will be sent to all staff. In addition, information regarding the research will be put on Trust and Nursing home websites and social media platforms e.g. Facebook and Twitter. Posters (appendix 8) will also be placed in communal areas ensuring information can be accessed by everyone. Staff will be directed to the researchers on the study via email or phone to discuss the study in more detail. For those who still wish to participate and who meet the inclusion criteria, written informed consent (appendix 7) will be obtained by the researcher(s).

Sample Collection: Once informed consent has been obtained each participant will provide (i) one 30 ml whole blood sample, one set of dried blood spots (DBS) and a saliva sample (~4ml) at recruitment. Then, only if SARS-CoV-2 symptoms such as a high temperature/a new continuous cough https://www.nhs.uk/conditions/coronavirus-covid-19/check-if-you-have-coronavirus-symptoms/ experienced during 2 week post recruitment period: (ii) a saliva sample, one 30 ml whole blood sample and one set of dried blood spots (DBS) and a lateral flow assay for COVID-19 antibodies performed (between 0 and 10 days of symptom onset), (iii) a saliva sample, one 30 ml whole blood sample and one set of DBS and a lateral flow assay for COVID-19 antibodies performed between 14-28 days after symptom onset (iii) a saliva sample, one extra set of 30ml whole blood and DBS to be taken only if pneumonia occurs during (usually only in severe symptom cases) (iv) In addition, where possible sample will also be collected at 3 months, 6 months and 12 months of symptom onset. Sample collections will take place at an agreed convenient time and place.

Data Collection for all cohorts (including COVRES2 follow up):

The phenomic data collected will align with international/National data for phenotypic data collection (HDRUK). After informed consent (appendices 3, 5 & 7) is obtained by a member of the research team, participants will be asked to answer a health and lifestyle questionnaire at each timepoint (Appendix 9) that includes questions about their general medical and clinical history such as comorbidities, medications, respiratory illness, COVID-19 symptomatology, time to admission to hospital (if hospitalised) as well as lifestyle habits, family history etc.

Missing information will be collected by the researchers by accessing the participants electronic care records or the participants medical notes provided concent has been obtained for this option. Demographic variables in addition to age and gender will include height, weight and blood pressure will also be retrieved from the participants electronic care record. The researchers will have an honorary contract within the Health Trust(s) and will have approval and training to access and to use the patient care records. In case certain information is missing, the researchers will ask permission to follow up with the patient at a later time by phone. All medical records will be accessed on the Altnagelvin hospital site at C-TRIC and information will be manually inputted to a database on a university password protected and encrypted laptop.

Participants will also be asked whether consent is cnfirmed at each time point, to complete a validated mental health questionnaire, the General Health Questionnaire (GHQ-12), (appendix 10) to assess the association between their condition or perceived risk and their mental health and wellbeing. The researchers will arrange for completion of this questionnaire at a convenient time for the participant either on the day of recruitment, during the follow up visits, online or by phone.

Participants also have the choice to consent to be contacted again to receive information regarding future studies.

Sample processing, storage and analysis

Saliva ~ 4ml will be collected in Oragene saliva collection kits (DNA Genotek), processed and analysed for COVID-19 genome sequencing and microbiome analysis.

Whole blood samples will be processed to extract plasma and flow cytometry. Paper discs will be punched out of dried blood spot samples (DBS) and protein, prescribed medication, drug metabolites and DNA extracted by addition of a routine elution buffer. Lateral flow data will be logged at the time at of assay and where possible dedicated COVID-19 app photograph of test strip result archived. DBS extracts and plasma samples will be logged, aliquoted and labelled with unique bar code identifiers prior to storage at -80'C in the Northern Ireland Centre for Stratified Medicine (NICSM) until analysis. DBS protein (IgG, C-reactive protein and cytokines and plasma will be analysed using ELISA and OLINK or drug metabolites by mass spectrometry. With participant agreement, DNA extracted from DBS/blood samples for future whole genome sequencing (WGS) and extracted drug metabolites will be stored at -80C in. A whole genome sequence will be generated from each participant DNA sample. A selected cohort of patient samples will also be subjected to transcriptomics (RNA Seq), microbiome and methylation analyses.

Whole blood samples and swab extract will undergo viral genome analyses sequencing, transcriptomics, epigenetics, single nucleotide polymorphism (SNP) genotyping, WGS and RNAseq generation. Sample analysis will be performed at NICSM by the researchers or by a third party such as the virology laboratories at Queens University Belfast (QUB), Regional Virus Laboratory Belfast (RVL), Olink® proteomics (Uppsala, Sweden) or Genomics Medicine Ireland (GMI, Dublin, Dublin). This will require aliquots of plasma/serum or DNA to be transferred to the approved third party proteomic or genomic or service providers (such as QUB, Olink or GMI). In this event, all samples will be pseudo-anonymised. The codes relating to participant identification will not be disclosed to this study partner and remain in the custody of the chief investigator. Third party providers have already been approved as service providers with satisfactory evidence of encryption in storage and transfer of data and appropriate Material Transfer, Confidentiality and Intellectual Property agreements signed off by both the third party and the University. Unused DNA or plasma which is analysed by a third party such as GMI or Olink® proteomics will be destroyed. The research organisations that will use samples or data derived from analysis of samples could be not-for-profit e.g. universities or for-profit commercial companies (such GMI). GMI, however, have agreed to undertake: SNP genotyping, WGS and RNAseq generation analysis at no cost. Participant's name, address and personal details will not be made available to any organisation beyond the study team

Analysis

All sequencing, methylation and proteoomic analysis out sourced to Azenta (GeneWiz), Genuity and Olink Proteomics. Flow cytometry and 16s microbiome analysis will be completed at CTRIC.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male and female
* Age: >18
* BMI: Any
* Ethnic origin: Any

Hospitalised, non-hospitalised and nursing home patients:

* Symptomatic/non-Symptomatic patients testing positive or suspected of being positive for COVID-19/SARS-CoV-2 by virus PCR assay
* Nursing homes caring for elderly residents
* COVID-19 wards of participating hospitals

Hospital and nursing home staff:

• Any member of primary care, hospital or nursing home staff (including GP's) are eligible to participate whether have ever tested positive or not for COVID- 19/SARS-CoV-2 by virus PCR assay even if non-symptomatic.

Exclusion Criteria:

All cohorts:

* Under 18 years of age
* Those with intellectual disabilities or mental health illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cohorts where recruited from the Western Health and Social Care Trust, Northern Ireland.
Sampling Method: Non-Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Hospitalisation severity status | 1 month
  Hospitalised and non hospitalied Covid-19 patients will be recruited onto the study for plasma and saliva biomarker assessment
Persistence of Covid-19 symptoms | 6 months
  Determination of whether Covid-19 symptoms have changed at 3 and 6 months

SECONDARY OUTCOMES:
Immunological assessment | 6 months
  To measure IgG to SARS-CoV-2 in a representative sample of the NI population at community level (nursing home), in hospitalised and non-hospitalised SARS-CoV-2 positive cases and in frontline healthcare staff (including GP's, primary care staff, hospital and nursing home staff).
Genomic assessment | 6 months
  To perform whole genome sequencing on phlebotomy blood samples from hospitalised SARS-CoV-2 positive cases and frontline healthcare staff who have received a SARS-CoV-2 vaccine and /or positive or negative for SARS-CoV-2 (including as above a.) and collect associated SARS-CoV-2 PCR test data, comorbidity and medication data.
Flow cytometry asessment of immune cells | 6 months
  To analyse immune cell and inflammatory responses in hospitalised and non-hospitalised SARS-CoV-2 positive cases and frontline healthcare staff who have received a SARS-CoV-2 vaccine and /or positive or negative for SARS-CoV-2 (including as above a.).

CONTACTS AND LOCATIONS:
Overall Officials: David Gibson, PhD, Principal Investigator — University of Ulster
Locations (1):
- Personalised Medicine Centre, School of Medicine, Ulster University, C-TRIC Building,, Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Discussions can be had on individual basis, to share data if requested.

REFERENCES:
- [Background] Merad M, Martin JC. Pathological inflammation in patients with COVID-19: a key role for monocytes and macrophages. Nat Rev Immunol. 2020 Jun;20(6):355-362. doi: 10.1038/s41577-020-0331-4. Epub 2020 May 6. PMID 32376901
- [Background] Moons KG, Altman DG, Reitsma JB, Ioannidis JP, Macaskill P, Steyerberg EW, Vickers AJ, Ransohoff DF, Collins GS. Transparent Reporting of a multivariable prediction model for Individual Prognosis or Diagnosis (TRIPOD): explanation and elaboration. Ann Intern Med. 2015 Jan 6;162(1):W1-73. doi: 10.7326/M14-0698. PMID 25560730
- [Background] Ong EZ, Chan YFZ, Leong WY, Lee NMY, Kalimuddin S, Haja Mohideen SM, Chan KS, Tan AT, Bertoletti A, Ooi EE, Low JGH. A Dynamic Immune Response Shapes COVID-19 Progression. Cell Host Microbe. 2020 Jun 10;27(6):879-882.e2. doi: 10.1016/j.chom.2020.03.021. Epub 2020 Apr 30. PMID 32359396
- [Background] Sun X, Wang T, Cai D, Hu Z, Chen J, Liao H, Zhi L, Wei H, Zhang Z, Qiu Y, Wang J, Wang A. Cytokine storm intervention in the early stages of COVID-19 pneumonia. Cytokine Growth Factor Rev. 2020 Jun;53:38-42. doi: 10.1016/j.cytogfr.2020.04.002. Epub 2020 Apr 25. PMID 32360420
- [Background] Tay MZ, Poh CM, Renia L, MacAry PA, Ng LFP. The trinity of COVID-19: immunity, inflammation and intervention. Nat Rev Immunol. 2020 Jun;20(6):363-374. doi: 10.1038/s41577-020-0311-8. Epub 2020 Apr 28. PMID 32346093
- [Background] Thevarajan I, Nguyen THO, Koutsakos M, Druce J, Caly L, van de Sandt CE, Jia X, Nicholson S, Catton M, Cowie B, Tong SYC, Lewin SR, Kedzierska K. Breadth of concomitant immune responses prior to patient recovery: a case report of non-severe COVID-19. Nat Med. 2020 Apr;26(4):453-455. doi: 10.1038/s41591-020-0819-2. No abstract available. PMID 32284614
- [Background] Vardhana SA, Wolchok JD. The many faces of the anti-COVID immune response. J Exp Med. 2020 Jun 1;217(6):e20200678. doi: 10.1084/jem.20200678. PMID 32353870
- See also: Penny Ward. COVID-19/SARS-CoV-2 Pandemic 2020.https://www.fpm.org.uk/blog/covid-19-sars-cov-2-pandemic/ — https://www.hdruk.ac.uk/projects/national-phenomics-resource/

DOCUMENTS (2):
  • Study Protocol (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT05548829/Prot_000.pdf
  • Informed Consent Form (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT05548829/ICF_001.pdf